CLINICAL TRIAL: NCT05328115
Title: A Double-blind, Randomized, Parallel-group Multiple Dose Study on the Safety, Tolerability and Immunogenicity of ALZ-101 in Participants With Early Alzheimer's Disease
Brief Title: A Study on the Safety, Tolerability and Immunogenicity of ALZ-101 in Participants With Early Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alzinova AB (Industry)
Collaborators: CRST Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALZ-C-001; 2019-002277-62 (EudraCT Number)
Record Dates: First submitted 2022-03-25; First posted 2022-04-14 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease; Dementia Alzheimers; Dementia, Mild
MeSH Terms: conditions — Alzheimer Disease; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The arm with ALZ-101 400 μg will be open-labelled treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ALZ-101 125 μg (Active Comparator): Intramuscular injection of 125 μg of ALZ-101 adjuvanted vaccine dosed once a month at four doses
  Interventions: Biological: ALZ-101
- ALZ-101 250 μg (Active Comparator): Intramuscular injection of 250 μg of ALZ-101 adjuvanted vaccine dosed once a month at four doses
  Interventions: Biological: ALZ-101
- Placebo (Placebo Comparator): Intamuscular Saline solution mixed adjuvant and dosed once a month at four doses
  Interventions: Other: Placebo
- ALZ-101 400 μg (Active Comparator): Intramuscular injection of 400 μg of ALZ-101 adjuvanted vaccine dosed once a month at four doses
  Interventions: Biological: ALZ-101

INTERVENTIONS:
Biological: ALZ-101 — Intramuscular injections of adjuvanted peptide vaccine against oligomeric Amyloid Beta.
  Arms: ALZ-101 125 μg; ALZ-101 250 μg; ALZ-101 400 μg
Other: Placebo — Intramuscular injections of adjuvanted placebo.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate safety, tolerability and immunogenicity of the vaccine ALZ-101 against Alzheimer's Disease. Patients diagnosed with early Alzheimer's will be included. The study have two parts. The Part A (including A1 and A2), includes four doses of ALZ-101 or corresponding placebo given over 16 weeks. Participant will be followed up to Week 30 in Part A1 and either continue in the extension part of the study, Part B, or complete Part A1. Participant not eligible to Part B will be followed up until Week 68 with no further dosing. Participant eligible for Part B will be treated with 2 doses of open-label ALZ-101, over 16 weeks and followed up during in total 68 weeks (Part A1 and B). Part A2 participants will be followed over 20 weeks.

ELIGIBILITY:
Main inclusion criteria in Part A:

1. Male and female subjects between 50 and 83 years (inclusive) of age at the time of informed consent
2. Subjects capable of providing valid independent informed consent and signing the informed consent form (the subjects' capacity to provide valid consent should be determined in accordance with applicable professional standards, and will be based on the Investigator's judgement)
3. Subjects with MCI due to AD or mild AD according to National Institute of Aging - Alzheimer's Association (NIA-AA) core clinical criteria; subjects must have all of the following at screening:

   1. CDR global score (GS) of 0.5 or 1
   2. CDR memory score of ≥0.5
   3. MMSE score of ≥20 points
4. Screening CSF results showing a pattern consistent with amyloid plaque load and indicative of AD pathology. The CSF results will be evaluated by the Investigator and will take into account the Aβ42/40 ratio (cut-off level set by the laboratory)
5. If the subject is receiving an acetylcholine esterase inhibitor (AChEI) or memantine or both for the treatment of MCI or AD, this treatment must be on a stable dosage for at least 8 weeks prior to the first dosing of IMP. Treatment-naïve subjects may also be entered into the study
6. Subjects must have an identified, reliable and knowledgeable study partner who is willing and able to support the participant and to provide follow-up information on the study participant throughout the course of the study. This person must, in the opinion of the Investigator, spend sufficient time with the study participant on a regular basis such that he or she can reliably fulfil the requirements of being a study partner (however, a study partner does not need to be living in the same household with the study participant)

Main inclusion criteria in Part B:

1. Male and female subjects who have completed Visit 15 of Part A and are willing to continue in Part B of the study
2. Subjects providing informed consent and signing the informed consent form. In case a subject is considered not to be capable of providing valid independent informed consent, the subject's legally acceptable representative (LAR) should consent to the study on behalf of the subject. In such a case, the subject should provide informed assent to continue in the study
3. Subjects must have an identified, reliable and knowledgeable study partner who is willing and able to support the participant and to provide follow-up information on the study participant throughout the course of the study. This person must, in the opinion of the Investigator, spend sufficient time with the study participant on a regular basis such that he or she can reliably fulfil the requirements of being a study partner.

Main exclusion criteria in Part A:

1. Subjects having any contraindication to MRI scanning; or are unable to undergo brain MRI scanning according to the standard criteria of the MRI unit; or the Investigator believes that the subject will not be able to undergo further scans scheduled during the course of the study
2. Screening MRI (3T) results showing evidence of clinically significant pathological lesions that could indicate a dementia-associated diagnosis other than early AD or cause a safety risk for the participant (a list of possible exclusionary findings is included in the main protocol text)
3. Modified Hachinski Ischemia Score (mHIS) >4 at screening
4. History of a cerebrovascular incident, including transient ischemic attack (TIA) or stroke, within 12 months of screening
5. Subject with a history of seizures within 2 years of screening
6. Any psychiatric diagnosis or symptoms (e.g. hallucinations, major depression, delusions, schizophrenia, bipolar disorder) that, in the opinion of the Investigator, could interfere with study procedures or assessments or participant safety. A subject with depression may, however, be included if treated with a stable dose of antidepressants for at least 8 weeks before screening and not fulfilling DSM-5 criteria for major depression at screening
7. Significant risk of suicide (defined using the Columbia Suicide Severity Scale [C-SSRS], with the subject answering "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behaviour) within 12 months of screening
8. Disorder related to alcohol or drug abuse, as defined in DSM-5, within 2 years prior to screening
9. Evidence of current or history of any significant autoimmune disease that, in the opinion of the Investigator, could interfere with evaluation of the study results or constitute a health hazard for the subject
10. Evidence of an immune system that is compromised; including, but not limited to, a diagnosis of HIV (human immunodeficiency virus); or the subject has been splenectomised or has received an organ transplant (corneal transplants excluded), or is receiving chronic systemic immunosuppressive medication
11. Evidence of current clinically significant and possibly unstable pulmonary, gastrointestinal, renal, hepatic, endocrine, hematological or cardiovascular system disease or metabolic disturbance
12. Diagnosis of cancer (hematological or solid tumor) for which the subject is currently being treated, or for which there has been treatment within 5 years preceding screening, or for which there is still evidence of active disease. Subjects with local prostate cancer or local dermatological tumors, such as basal or squamous cell carcinoma, may be included
13. Any clinically significant abnormalities in laboratory tests, vital signs, ECG or physical examination findings at screening that in the opinion of the Investigator require further investigation or treatment, or may interfere with study procedures or safety. These may include, but are not limited to, the following:

    1. estimated glomerular filtration ratio (eGFR) <30 ml/min/1.73 m2, based on the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation
    2. plasma total bilirubin value >2 times the upper limit of the reference range
    3. plasma alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) value >2 times the upper limit of the reference range
    4. low vitamin B12 or folate values that are considered to be clinically significant in relation to cognitive impairment. In such cases, re-screening is permissible after supplementation therapy has been provided for a sufficient time
    5. prolonged QTcF interval of >470 ms
14. Clinically suspected active neuroborreliosis, confirmed by the presence of Borrelia antibodies in CSF
15. Contraindication to lumbar puncture (LP). These contraindications may include, but are not limited to, the following:

    1. increased intracranial pressure (ICP)
    2. skin infection at the LP site
    3. significant lumbar spine deformity
    4. bleeding diathesis (e.g., significant thrombocytopenia)
    5. taking anticoagulant therapy (e.g., warfarin, dabigatran, apixaban, or other blood factor or thrombin inhibitor). Use of anti-platelet therapy (e.g. low dose aspirin) may be permitted if deemed appropriate in the Investigator's judgement
16. Current or anticipated use, or recent prior use (pre-study time limits specified in the main protocol text) of disallowed concomitant treatment
17. Any vaccination within 2 weeks prior to screening
18. History of severe drug allergy (anaphylactic shock or drug-induced hypersensitivity syndrome), or known hypersensitivity to vaccines, including constituents of vaccines Having received in another clinical trial

    1. any therapeutic monoclonal antibody, protein derived from a monoclonal antibody or immunoglobulin therapy within 6 months before screening
    2. active anti-amyloid immunization or other active immunization for the treatment of AD
    3. any other investigational medication (unless it can be documented that the subject received only placebo) or device within 3 months or 5 half-lives (whichever is longer) before screening

20. Any condition that may be contributing to cognitive impairment above and beyond that caused by the subject's early AD 21. Disease or medication that, in the opinion of the Investigator, could interfere with the assessments of safety, tolerability or immunogenicity 22. Planned surgery that would take place during the double-blind treatment period of the study. Planned surgery not requiring general anaesthesia need not result in exclusion, if in the opinion of the Investigator this operation does not interfere with study procedures and participant safety 23. Blood donation or loss of significant amount of blood within 3 months prior to the first screening visit 24. Female subjects of childbearing potential

Main exclusion criteria in Part B:

1. Any new condition that may be contributing to cognitive impairment above and beyond that caused by the subject's AD
2. Any new disease or medication that, in the opinion of the Investigator, could interfere with the assessments of safety, tolerability or immunogenicity or constitute a health hazard for the subject participating in Part B of the study; however, a new disease or medication that would prevent CSF sample collection in Part B need not result in exclusion

Ages: 50 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) and serious AEs (SAEs) | From enrolment through study completion, an average 1 year
  Any adverse or serious adverse events that could be associated with the study procedure.
Number of participants with treatment-emergent AEs and SAEs | From enrolment through study completion, an average 1 year
  Any adverse or serious adverse events that could be associated with the treatment.
Number of AEs of special interest (AESIs), including injection-related events (IREs)and amyloid-related imaging abnormalities (ARIAs) | From enrolment through study completion, an average 1 year
  Any adverse or adverse events of special interest that could be associated with the treatment.
Number of participants with clinically significant cognitive or functional worsening of Alzheimer's Disease(AD) according to Alzheimer's DiseaseCooperative Study -Clinician's Global Impression of Change (ADCS-CGIC)scores of 6 and 7 | From first dose to study completion, an average 1 year
  Any clinically significant worsening of cognitive functions as assessed by Alzheimer's DiseaseCooperative Study -Clinician's Global Impression of Change [ADCS-CGIC]scores. Scores are graded from 1 to 7, where 1 means very much improved cognitive function and 7 very much worsening cognitive function.

SECONDARY OUTCOMES:
Aβ-specific antibody titre | From first dose to study completion, an average 1 year
  Aβ-specific antibody titre of post-baseline samples (if baseline sample is negative) OR titre fold increase defined as the ratio of any post-baseline Aβ-specific antibody titre to baseline antibody titre in serum
Number of titre-based responders | From first dose to study completion, an average 1 year
  Number of titre-based responders, defined as post-baseline sample becoming positive for Aβ-specific antibodies(if baseline sample is negative) OR post-baseline titre at least four times the baseline antibody titre in serum
Area under serum Aβ-specific antibody titre curve (AUC) | From first dose to week 20
  Area under serum Aβ-specific antibody titre curve (AUC) from Week 0 to Week 20.

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, MD, Principal Investigator — CRST Oy
Locations (1):
- Clinical Research Services Turku -CRST Oy, Turku, Finland

IPD SHARING:
Plan to Share IPD: No